CLINICAL TRIAL: NCT05904795
Title: Comparative Effects of Proprioceptive Neuromuscular Facilitation Strengthening Exercises and De-lorme and Watkins Exercises Program on Upper Limb Function and Strength in Chronic Stroke Patients
Brief Title: PNF Strengthening and De-lorme and Watkins Exercises on Upper Extremity Function and Strength in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/LHR/23/0215 ZAINAB TEHREEM
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Upper Extremity Paresis
Keywords: Proprioceptive neuromuscular facilitation
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF strengthening exercises (Active Comparator): Pnf strengthening exercises along with isometrics and range of motion exercises
  Interventions: Other: PNF strengthening exercises
- de-lorme and watkins progressive resistance exercises (Active Comparator): progressive resistance exercises along with isometrics and range of motion exercises
  Interventions: Other: de-lorme and watkins exercises

INTERVENTIONS:
Other: PNF strengthening exercises — PNF strengthening exercises 10 repetitions, 1set , 4 days/week along with range of motion exercises total of 4 sessions were given consisting 40 minutes
  Arms: PNF strengthening exercises
Other: de-lorme and watkins exercises — The group was given de-lorme and watkins progressive resistance exercises along with range of motion exercises .10 repetitions, 1set, 4 days /week along with range of motion exercises.
  total of 4 sessions per week each consisting of 40 minutes.
  Arms: de-lorme and watkins progressive resistance exercises

SUMMARY:
The aim of this study is to evaluate the effects of proprioceptive neuromuscular facilitation strengthening exercises and de-Lorme and Watkins exercises program in stroke patients with upper limb weakness in chronic stroke patients. The randomized central trial will recruit patients according to consecutive sampling into two intervention groups. One group will receive proprioceptive neuromuscular facilitation strengthening exercises and other group will receive de-Lorme and Watkins exercises program.

DETAILED DESCRIPTION:
A study in which the participants (n=26) were recruited in the study suffering from stroke and meeting the inclusion criteria. Two groups formed such that patients in group A will be treated with conventional therapy and PNF and group B will be treated with PNF and NMES in along with conventional therapy. The protocol will cover 6 weeks of treatment. Regular assessment at 0,3rd and 6th week will be carried out. In the rehabilitation period, we will evaluate upper extremity function, activities of daily living(ADLs), mental status examination at regular interval during the rehabilitation.In previous studies there is less literature regarding the combine effects of proprioceptive neuromuscular facilitation techniques and de-Lorme and Watkins exercise program on upper limb function and strength in chronic stroke patients with upper limb weakness. Therefore there is dire need to explore which training technique is most effective in improving upper limb function and strength in chronic stroke patients therefore this study aims in comparative effects of proprioceptive neuromuscular facilitation strengthening exercises and de-Lorme and Watkins exercise program on upper limb function and strength in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients.
* Medically stable patients having a single stroke.
* History of stroke 6 to 24 months.
* A score greater than 24-30 in mini-mental test.
* Patients having consciousness with GC;10

Exclusion Criteria:

* Recurrent stroke
* Patients with gullian berrie syndrome, multiple sclerosis lesion osteoarthritis of shoulder.
* Manual muscle testing below grade II.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The barthel index scale | 4th day
  The Barthel Index (BI) is a measure of independence in activities of daily living (ADL).It contains 10 components which has different scores.The total score is calculated by dividing 100.
Hand held dynamometer | 4th day
  The hand held dynamometry is an objective method in detecting minimum muscle strength change, which has an impact on the physical function of ICU survivors. The minimum change in the fore can be measured in units of weight such as pounds or kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, MSNMPT, Principal Investigator — Riphah International Universiry
Locations (1):
- Shahida Islam teaching hospital Lodhran, Lodhran, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade SE, Harrold LR, Tjia J, Cutrona SL, Saczynski JS, Dodd KS, Goldberg RJ, Gurwitz JH. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic attack using administrative data. Pharmacoepidemiol Drug Saf. 2012 Jan;21 Suppl 1(Suppl 1):100-28. doi: 10.1002/pds.2312. PMID 22262598
- [Background] Zuber M, Mas JL. [Epidemiology of cerebrovascular accidents]. Rev Neurol (Paris). 1992;148(4):243-55. French. PMID 1439451
- [Background] Gillespie CD, Wigington C, Hong Y; Centers for Disease Control and Prevention (CDC). Coronary heart disease and stroke deaths - United States, 2009. MMWR Suppl. 2013 Nov 22;62(3):157-60. PMID 24264507
- [Background] Mergenthaler P, Dirnagl U, Meisel A. Pathophysiology of stroke: lessons from animal models. Metab Brain Dis. 2004 Dec;19(3-4):151-67. doi: 10.1023/b:mebr.0000043966.46964.e6. PMID 15554412
- [Background] Harris JE, Eng JJ. Paretic upper-limb strength best explains arm activity in people with stroke. Phys Ther. 2007 Jan;87(1):88-97. doi: 10.2522/ptj.20060065. Epub 2006 Dec 19. PMID 17179441
- [Background] Hendricks HT, van Limbeek J, Geurts AC, Zwarts MJ. Motor recovery after stroke: a systematic review of the literature. Arch Phys Med Rehabil. 2002 Nov;83(11):1629-37. doi: 10.1053/apmr.2002.35473. PMID 12422337
- [Background] Pak S, Patten C. Strengthening to promote functional recovery poststroke: an evidence-based review. Top Stroke Rehabil. 2008 May-Jun;15(3):177-99. doi: 10.1310/tsr1503-177. PMID 18647724